CLINICAL TRIAL: NCT06471205
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of BL-B01D1+PD-1 Monoclonal Antibody Combination Therapy in Patients With Unresectable Locally Advanced or Recurrent Metastatic Triple-negative Breast Cancer
Brief Title: A Study of BL-B01D1+PD-1 Monoclonal Antibody in Patients With Unresectable Locally Advanced or Recurrent Metastatic Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-204-04
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1+PD-1 Monoclonal Antibody (Experimental): Participants receive BL-B01D1+PD-1 Monoclonal Antibody as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: PD-1 Monoclonal Antibody

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion on D1 and D8, or D1 for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: PD-1 Monoclonal Antibody — Administration by intravenous infusion for a cycle of 3 weeks (Q3W).

SUMMARY:
This phase II study is a clinical study to explore the efficacy and safety of BL-B01D1 combined with PD-1 monoclonal antibody in patients with unresectable locally advanced or recurrent metastatic triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. Age: ≥18 years old and ≤75 years old;
3. Expected survival time ≥3 months;
4. ECOG 0 or 1;
5. Subjects with histologically and/or cytologically confirmed, inoperable locally advanced or recurrent or metastatic triple-negative breast cancer;
6. Patients should not have received previous systemic therapy for unresectable, locally advanced, recurrent, or metastatic triple-negative breast cancer;
7. A archived tumor tissue specimen or fresh tissue specimen of the primary or metastatic lesion within 2 years must be provided;
8. Must have at least one place in accordance with RECIST v1.1 define measurable lesions;
9. No blood transfusion, no use of cell growth factors and/or platelet raising drugs within 14 days before screening, and the organ function level must meet the requirements;
10. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
11. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, the serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. ADC drugs that have received topoisomerase I inhibitors as small molecule toxins;
2. Palliative radiotherapy within 2 weeks before the first dose;
3. Patients with checkpoint inhibitors prior to neoadjuvant/adjuvant chemotherapy;
4. Use of an immunomodulatory drug within 14 days before the first dose of study drug;
5. The history of severe cardiovascular and cerebrovascular diseases in the past six months was screened;
6. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
7. Active autoimmune and inflammatory diseases;
8. Receiving long-term systemic corticosteroid therapy, etc., before the first dose;
9. Other malignant tumors that progressed or required treatment within 5 years before the first dose;
10. Presence of: a) poorly controlled diabetes mellitus before starting study treatment; b) severe complications associated with diabetes mellitus; c) a glycated hemoglobin level of 8% or more; d) hypertension poorly controlled by two antihypertensive drugs; e) history of hypertensive crisis or hypertensive encephalopathy;
11. Present grade ≥2 radiation pneumonitis according to the RTOG/EORTC definition; Patients with current ILD;
12. Complicated with pulmonary diseases leading to clinically severe respiratory impairment;
13. 6 months prior to screening needs treatment intervention unstable thrombotic events;
14. Patients with active central nervous system metastases;
15. Patients with massive or symptomatic effusions or poorly controlled effusions;
16. Allergic history to recombinant humanized antibody or human-mouse chimeric antibody or allergic to any excipients of the test drug;
17. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation;
18. HIV antibody positive, active tuberculosis, active hepatitis B virus infection, or active hepatitis C virus infection;
19. Serious infection within 4 weeks before the first dose of study drug; Signs of pulmonary infection or active pulmonary inflammation within 4 weeks;
20. Participated in another clinical trial within 4 weeks before the first dose;
21. Patients with superior vena cava syndrome should not be rehydrated;
22. Have a history of psychotropic substance abuse with an inability to quit or a history of severe neurological or psychiatric illness;
23. Imaging examination showed that the tumor had invaded or wrapped the large thoracic vessels;
24. Serious unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
25. Clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
26. Subjects who are scheduled to receive live vaccine or receive live vaccine within 28 days before the first dose;
27. Other circumstances considered by the investigator to be inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, Principal Investigator — Fudan University; Jian Zhang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China